CLINICAL TRIAL: NCT03361163
Title: Group A Streptococcal Human Challenge Study: Building a Pharyngitis Model to Accelerate Vaccine Development
Brief Title: Controlled Human Infection for Vaccination Against Streptococcus Pyogenes
Acronym: CHIVAS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Andrew Steer (Other)
Collaborators: University of Melbourne (Other); Nucleus Network Ltd (Other); National Health and Medical Research Council, Australia (Other); Telethon Kids Institute (Other); The Peter Doherty Institute for Infection and Immunity (Other); Queen Fabiola Children's University Hospital (Other); Griffith University (Other); University of Wollongong (Other); The University of Queensland (Other); University of Auckland, New Zealand (Other); University of Tennessee (Other)
Responsible Party: Sponsor-Investigator, Andrew Steer, Professor, Group A Streptococcal Research Group Leader, Murdoch Childrens Research Institute
Organization: Murdoch Childrens Research Institute (Other)
Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: CHIVAS-M75
Record Dates: First submitted 2017-11-14; First posted 2017-12-04 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Streptococcus Pyogenes Pharyngitis; Streptococcus Pharyngitis; Strep Throat; Streptococcus Pyogenes Infection; Group A Streptococcus: B Hemolytic Pharyngitis; Group A Streptococcal Infection; Gram-Positive Bacterial Infections; Bacterial Infections
Keywords: Streptococcus pyogenes pharyngitis; Streptococcus Pharyngitis; Strep Throat; Streptococcus pyogenes Infection; Group A Streptococcus: B Hemolytic Pharyngitis; Group A Streptococcal Infection; Controlled human infection model; Challenge study
MeSH Terms: conditions — Streptococcal Infections; Gram-Positive Bacterial Infections; Bacterial Infections

STUDY DESIGN:
Intervention Model Description: Observational, sequential, dose-escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GAS oropharyngeal challenge (Experimental): Biological: emm75 Streptococcus pyogenes (GAS M75, strain 611024)
  Direct oropharyngeal application using a sterile-tipped Dacron swab after immersion for 10 seconds in a 1mL vial containing 1-3x10^4 to 1-3x10^8 colony forming units (CFU) of the challenge strain (depending on dose group allocation).
  Interventions: Biological: emm75 Streptococcus pyogenes (GAS M75, strain 611024)

INTERVENTIONS:
Biological: emm75 Streptococcus pyogenes (GAS M75, strain 611024) — Direct oropharyngeal application by swab following immersion in a solution containing a specified concentration (dose) of GAS M75.
  Other Names: GAS M75; Group A Streptococcus challenge inoculum

SUMMARY:
Group A Streptococcus (GAS) infection is a major cause of death and disability globally with a disproportionately high burden in settings of disadvantage worldwide. Acute infections due to GAS range from very common superficial skin infections (>150 million prevalent cases) and pharyngitis (over 600 million incident cases) to life-threatening invasive disease (>600,000 incident cases) such as necrotising fasciitis. Post-infectious GAS sequelae of GAS include acute rheumatic fever (ARF, ~500,000 incident cases) leading to rheumatic heart disease (RHD, ~34 million prevalent cases), and acute glomerulonephritis. The health services impact of GAS disease in all its forms is immense and strikes at every level from primary to intensive care.

Controlled human infection models (CHIMs) have a long history of critical contributions to vaccine development. Data from CHIMs meeting modern scientific, regulatory, and ethical standards, are aiding efforts to control over 25 major human pathogens, including bacteria (e.g. pneumococcus, cholera), viruses (e.g. respiratory syncytial virus, influenza), and parasites (e.g. malaria, schistosomiasis).

A reliable and safe controlled human infection model of GAS pharyngitis will be an important part of the global vaccine development effort. To build the model, the investigators are undertaking a dose-ranging study using an observational, dose-escalation, inpatient trial to determine the dose of GAS administered by direct oropharyngeal inoculation (bacteria 'painted' onto throat) required to reliably produce a pharyngitis attack rate of ≥ 60% in carefully screened healthy adult volunteers.

DETAILED DESCRIPTION:
Group A Streptococcus (GAS) is a ubiquitous human pathogen. Its impact begins in early childhood and is felt most by those who have the least. Globally, the health services impact of GAS disease in all its forms is immense and strikes at every level from primary to intensive care. Despite recognition of the need for GAS vaccine development, there are major obstacles impeding progress. A human challenge model promises to help to shift inertia in GAS vaccine development.

The objective of this study is to use an observational, dose-escalation, inpatient trial to determine the dose of GAS administered by direct oropharyngeal inoculation required to reliably produce a pharyngitis attack rate of ≥ 60% in carefully screened healthy adult volunteers. A GAS strain has been specially selected and prepared for this study to ensure safety and clinical relevance. Potential participants aged 18 to 40 years, the age range associated with the lowest risk of invasive GAS disease, will be carefully screened to minimise risk and maximise the likelihood of achieving the pharyngitis endpoint.

The results of three human GAS pharyngeal vaccine-challenge studies from the 1970s are encouraging, and reassuring. GAS challenge did cause pharyngitis and was safe, with all participants responding to antibiotics and none experiencing complications, despite these studies using more aggressive GAS strains.

The study design involves direct oropharyngeal inoculation of GAS to sequential cohorts. Up to four doses will be tested, from 1-3 x 10^5 cfu/mL (lower than previous GAS challenge studies) to a maximum of 1-3 x 10^8 cfu/mL. A minimum of 20 and maximum of 80 participants will be challenged. The challenge procedure aligns closely that used successfully in the 1970s GAS human challenge studies. An incubation period of 36 to 72 hours is expected before onset of symptoms. Participants will be intensively monitored inpatients for up to six days after challenge. The primary outcome measure is GAS pharyngitis, as defined by a combination of positive clinical and laboratory features. All participants developing pharyngitis will be treated with antibiotics and and those without pharyngitis will also be treated after 5 days. Participants will be followed as outpatients at 1 week, and 1, 3, and 6 months after discharge.

*Due to an unexpectedly very high proportion of participants developing pharyngitis at the starting dose, scope for dose de-escalation was subsequently included in a protocol amendment, using a dose of 1-3 x 10^4 cfu/mL.

A challenge model also promises an unprecedented opportunity to use modern techniques to describe the immunobiology of GAS infection. Blood and saliva samples will be collected at multiple timepoints before, during, and after the challenge. Testing of serial samples will add a dynamic next level to the clinical foundations of the challenge model, enabling in-depth comparison between participants developing pharyngitis or not and paving the way to identifying immune correlates of protection.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, aged 18 - 40 years (inclusive) on the day of informed consent.
* Medically healthy, determined by medical history, physical examination, transthoracic echocardiogram, non-clinically significant laboratory profiles, vital signs, and 12-lead ECG at screening, as deemed by the investigator.
* No active or chronic diseases/disorders, no history of hospitalisation for illness within the six months prior to enrolment into study, and no major surgery within the 12 months prior to enrolment into study.
* Body mass index of 18.0 - 32.0 kg/m2 and body weight ≥ 50.0kg
* Systolic blood pressure (SBP) of 90 mmHg - 140 mmHg and diastolic blood pressure (DBP) of 50 mmHg - 90 mmHg. Vital signs can be repeated up to two times.
* Resting heart rate (HR), as measured by ECG of 40bpm - 100 bpm (confirmed by one repeat at screening).
* Females must be non-pregnant, non-lactating or postmenopausal for at least 1 year (as confirmed by follicle-stimulating hormone [FSH]), or surgically sterile for at least 6 months prior to dosing.
* All male and females of childbearing potential must agree to use two forms of acceptable contraception from the time of signing informed consent until 30 days after final dose of rifampicin.
* Acceptable forms of contraception include: barrier method (eg. condom, diaphragm); pharmacological hormonal methods (oral contraceptive pill, long-acting implantable, intrauterine device).
* Rifampicin may reduce the activity of oral and implantable contraceptives (not intrauterine devices) so additional use of a barrier method is required for 30 days after the final dose of rifampicin for participants using these methods.
* Participants who abstain from penile-vaginal intercourse are eligible when this is their preferred and usual lifestyle. These participants must not be planning in vitro fertilization within the study and follow-up period.
* Must be willing and able to read, understand, and sign the participant information and consent form.
* Able and willing (in the Investigator's opinion) to comply with all study requirements, including the in-patient confinement period and outpatient visits for the duration of the study (approximately 6 months including follow-up visits).

Exclusion Criteria:

* History of any clinically important cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, and renal, or other major disease, as determined by the Investigator.
* History of tonsillectomy, adenoidectomy or splenectomy.
* Known or suspected autoimmune disease or impairment/alteration of immune function resulting from:
* Congenital or acquired immunodeficiency (including immunoglobulin A deficiency)
* Receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months.
* Presence or history of a severe drug hypersensitivity, or allergic disease diagnosed and treated by a physician or history of a severe allergic reaction, anaphylaxis or convulsions following any vaccination or infusion.
* Personal or family history of severe GAS infection or sequelae (such as acute rheumatic fever, rheumatic heart disease, post-streptococcal glomerulonephritis) or invasive GAS disease (toxic shock syndrome, necrotizing fasciitis, bloodstream infection, pleural empyema, meningitis).
* Clinically significant disease or any condition or disease that might affect drug absorption, distribution or excretion, e.g. gastrectomy, diarrhea.
* Any vaccination within the last 28 days or use of any antibiotic therapy during the 14 days before challenge.
* Presence of acute infectious disease or febrile illness (e.g., sub-lingual temperature ≥ 38.5°C) within the five days prior to inoculation.
* Significant acute or chronic infection within 14 days prior to inoculation that the Investigator deems may compromise participant safety.
* Any clinically significant abnormal finding on biochemistry or haematology blood tests, urine analysis, ECG or transthoracic echocardiogram.
* Positive serologic results for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibodies.
* Ex-smoker with a >10 pack year smoking history or a current smoker who is unable to stop smoking for the duration of the study
* History or presence of alcohol abuse (defined as regular alcohol consumption of more than 40g per day) or drug habituation, or any prior intravenous usage of an illicit substance.
* A positive urine drug test at screening or admission for confinement (e.g., amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, and opiates) unless there is an explanation acceptable to the investigator or sub-investigator (e.g. the participant has stated in advance that they consumed a prescription or over-the-counter product which contained the detected drug) and the participant has a negative urine drug screen on retest.
* A positive alcohol breath test at screening or admission for confinement.
* Known hypersensitivity or other contraindication to use of penicillin, rifampicin or any other beta-lactam or rifamycin antibiotic(s).
* Known hypersensitivity or contraindication to both azithromycin and clindamycin.
* Known hypersensitivity to soya protein.
* Intolerance of throat swab procedure (exaggerated gag reflex).
* Any systemic corticosteroid (or equivalent) treatment in the 14 days prior to challenge, or for more than seven consecutive days within the past 3 months.
* Any corticosteroids, anti-inflammatory drugs (besides sporadic use of non-steroidal anti-inflammatory drugs), immunomodulators or anticoagulants in the previous 3 months, or anticipated use of such drugs during the study period. Any participant currently receiving or having previously received immunosuppressive therapy, including systemic steroids including adrenocorticotrophic hormone (ACTH) or inhaled steroids in dosages which are associated with hypothalamic-pituitary-adrenal axis suppression such as 1 mg/kg/day of prednisone or its equivalent or chronic use of inhaled high potency corticosteroids (budesonide 800 μg or fluticasone 750 μg per day). Intranasal corticosteroid use is not allowed from 14 days prior to admission, during the confinement period, and is discouraged prior to the first outpatient visit. Topical corticosteroid use is allowed.
* Use of prescription or non-prescription drugs and herbal supplements (such as St John´s Wort) within 14 days or 5 half-lives (whichever is the longer) prior to the inoculation administration. Use of vitamin supplements taken at standard doses is allowed.
* Participation in a research study that involved blood sampling of more than 450 mL/unit of blood, received or donated blood, blood products and/or plasma derivatives or any parenteral immunoglobulin preparation within 3 months of informed consent.
* History of severe infectious disease requiring hospitalisation for intravenous antibiotics.
* History of cancer (except adequately treated squamous cell or basal cell carcinoma of the skin and cervical intraepithelial neoplasia).
* Presence of implants or prosthesis (e.g. artificial joints, pacemakers).
* Participation in another research study within the 30 days prior to enrolment involving an investigational product or other intervention that might affect risk of invasive GAS infection or compromise the integrity of the study (e.g. significant volumes of blood already taken in previous study).
* Any significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the results of the study, or the participant's ability to participate in the study.
* Any employee of the sponsor or research site personnel directly affiliated with this study or their immediate family members defined as a spouse, parent, sibling, or child whether biological or legally adopted.
* Evidence of pre-existing immunity to the challenge strain as determined by quantitative +/- functional antibody testing of serum collected at the screening visit

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-09-28 (Actual); Study Completion 2020-04-21 (Actual)

PRIMARY OUTCOMES:
Proportion of participants at each GAS M75 dose level meeting the study pharyngitis endpoint | Up to 6 days after challenge dose administered.
  Proportion of participants at each GAS M75 dose level who develop pharyngitis, using a combined clinical-microbiological definition comprising sore throat, physical examination signs of pharyngitis and tonsillitis, and microbiological confirmation of GAS by culture and nucleic acid amplification test of throat swabs.

CONTACTS AND LOCATIONS:
Overall Officials: Janet Wong, MBBS,BSc, Principal Investigator — Senior Medical Officer, Nucleus Network Limited; Andrew C Steer, MBBS,MPH,PhD, Principal Investigator — Group A Streptococcal Research Group, Murdoch Children's Research Institute
Locations (1):
- Centre for Clinical Studies (Nucleus Network Limited), Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Osowicki J, Azzopardi KI, Fabri L, Frost HR, Rivera-Hernandez T, Neeland MR, Whitcombe AL, Grobler A, Gutman SJ, Baker C, Wong JMF, Lickliter JD, Waddington CS, Pandey M, Schuster T, Cheng AC, Pollard AJ, McCarthy JS, Good MF, Dale JB, Batzloff M, Moreland NJ, Walker MJ, Carapetis JR, Smeesters PR, Steer AC. A controlled human infection model of Streptococcus pyogenes pharyngitis (CHIVAS-M75): an observational, dose-finding study. Lancet Microbe. 2021 Jul;2(7):e291-e299. doi: 10.1016/S2666-5247(20)30240-8. Epub 2021 Apr 15. PMID 35544165
- [Derived] Fabri LV, Azzopardi KI, Osowicki J, Frost HR, Smeesters PR, Steer AC. An emm-type specific qPCR to track bacterial load during experimental human Streptococcus pyogenes pharyngitis. BMC Infect Dis. 2021 May 21;21(1):463. doi: 10.1186/s12879-021-06173-w. PMID 34020607
- [Derived] Osowicki J, Azzopardi KI, Baker C, Waddington CS, Pandey M, Schuster T, Grobler A, Cheng AC, Pollard AJ, McCarthy JS, Good MF, Walker MJ, Dale JB, Batzloff MR, Carapetis JR, Smeesters PR, Steer AC. Controlled human infection for vaccination against Streptococcus pyogenes (CHIVAS): Establishing a group A Streptococcus pharyngitis human infection study. Vaccine. 2019 Jun 6;37(26):3485-3494. doi: 10.1016/j.vaccine.2019.03.059. Epub 2019 May 14. PMID 31101422